CLINICAL TRIAL: NCT04593316
Title: Study of Risk Factors for the Occurrence and Severity of Exertional Heatstroke in the Military Environment
Acronym: EXPLO-CCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PBMD03; 2020-A01967-32 (Other: IDRCB)
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Heat Stroke
MeSH Terms: conditions — Heat Stroke | interventions — Surveys and Questionnaires; Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exertional heatstroke group: Patients presenting or having presented exertional heatstroke.
  Interventions: Other: Saliva collection; Behavioral: Questionnaires; Other: Ingestible core temperature capsule intake; Other: Physical exercise; Other: Heart rate monitoring; Other: Core temperature monitoring
- Control group: Healthy people who never experienced exertional heatstroke.
  Interventions: Other: Saliva collection; Behavioral: Questionnaires; Other: Ingestible core temperature capsule intake; Other: Physical exercise; Other: Heart rate monitoring; Other: Core temperature monitoring

INTERVENTIONS:
Other: Saliva collection — A saliva sample will be collected before physical exercise.
Behavioral: Questionnaires — The participant will fill in questionnaires relative to his heath status and psychological and motivational resource questionnaires before physical exercise.
Other: Ingestible core temperature capsule intake — The participant will ingest a capsule before physical exercise in order to continuously monitor core temperature during physical exercise.
Other: Physical exercise — The participant will perform a walk/run test.
Other: Heart rate monitoring — Heart rate will be monitored during physical exercise thanks to a chest belt.
Other: Core temperature monitoring — Heart rate will be monitored during physical exercise thanks to an ingestible core temperature capsule.

SUMMARY:
Although the circumstances of onset and management of exertional heatstroke have been identified for several years, its pathophysiology remains imperfectly understood. Exertional heatstroke is the result of both extrinsic (i.e. environmental) and intrinsic (i.e. individual) contributing factors.

Extrinsic factors are well known (high ambient temperature and hygrometry, poorly "breathable" clothing, intense and prolonged physical effort) but some of them may be observed in milder conditions. In the French Armed Forces, 25% of the exertional heatstrokes that have been reported between 2005 and 2011 occurred below 17°C.

Intrinsic factors, on the other hand, are numerous and less consensual, partly because of the imperfect knowledge of exertional heatstroke physiopathology. Potential factors include a thermoregulatory defect (inability to maintain a temperature plateau during an effort) and several genetic mutations may also contribute to explain a propensity to present an exertional heatstroke. While exertional heatstroke is clearly not a monogenic pathology, the association of several polymorphisms could contribute to this vulnerability. Among the genes that have been explored, mutations in ryanodine receptor type 1 (RyR 1), calsequestrin-1 or angiotensin-1 converting enzyme (ACE) appear to be potential candidates. However, it is very likely that other polymorphisms may be involved, such as: genes involved in sports performance and exercise rhabdomyolysis, in the inflammatory cascade, permeability of the digestive epithelial barrier, adenosine receptors and susceptibility to anxiety.

Finally, motivation is a mixed factor often claimed to be involved in exertional heatstroke but has never been quantified and needs to be objectified.

To date, none of these hypotheses has been clearly assessed by comparing patients who experienced exertional heatstroke to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Active military
* Between 18 and 45 years old
* Ability to the walk/run test

Exclusion Criteria:

* Ongoing drug treatment (for the control group only),
* BMI greater than or equal to 30,
* Contraindication to the ingestion of a core temperature capsule

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be composed of patients who are experiencing or who have experienced exertional heatstroke (heatstroke group) and people who have not (control group).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Difference of the frequency of CYP24A1 gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of CYP24A1 gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of DRD2 gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of DRD2 gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of BDNF gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of BDNF gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of COMT gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of COMT gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of FAAH gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of FAAH gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of TPH2 gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of TPH2 gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of GRIN2B gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of GRIN2B gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of PER3 gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of PER3 gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of TNF-a gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of TNF-a gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of IL-6 gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of IL-6 gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of IL1B gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of IL1B gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of HSPA1B gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of HSPA1B gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.
Difference of the frequency of TLR4 gene polymorphisms between the heatstroke group and the control group | At enrollment (day 1)
  The frequency of TLR4 gene polymorphisms will calculated in each group by dividing the number of participants who present the polymorphism by the total number of participants in the group.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge
  - Hôpital d'Instruction des Armées Laveran, Marseille
  - Ecole du Val-de-Grâce, Paris